CLINICAL TRIAL: NCT07004478
Title: Turkish Adaptation, Validity and Reliability Study of the Generic Functional Index
Brief Title: Turkish Adaptation Study of the Generic Functional Index
Status: Recruiting | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Other Study IDs: IstanbulBUFC9
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Diseases
Keywords: function; musculoskeletal; reliability; validity; Generic Functional Index
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with musculoskeletal conditions: The sample will include adult individuals presenting with various musculoskeletal disorders, including but not limited to low back pain, osteoarthritis, tendinopathies, or other soft tissue conditions, which may influence their functional status.
  Interventions: Other: Translating the Generic Functional Index into Turkish and Related Processes; Other: Validity; Other: Internal consistency and Reliability

INTERVENTIONS:
Other: Translating the Generic Functional Index into Turkish and Related Processes — The translation process will follow a specific protocol in accordance with the guidelines. It will include two independent forward translations and one back-translation, conducted after obtaining written permission from the original authors. Discrepancies between translations will be reviewed by an expert committee to resolve terminological and cultural differences. The process will ensure conceptual and cultural equivalence between the original English version and the Turkish version. The final version of the questionnaire will be adapted to the target population and finalized in consultation with the original authors.
Other: Validity — Content validity will be calculated with the Content Validity Index, which is a result of expert opinions in terms of clarity, difficulty, and suitability of the Turkish version of the Generic Functional Index.
Other: Internal consistency and Reliability — The internal consistency of the items will be tested with Cronbach alpha. Test-retest reliability will be tested with intraclass correlation coefficient.

SUMMARY:
The Generic Functional Index is a scale developed to assess the general functional status of individuals. This study aims to evaluate the validity and reliability of the Turkish version of the Generic Functional Index. The adaptation process was designed to follow a standardized translation protocol, including forward translation, expert committee review, back-translation, pilot testing, and psychometric analyses. Data will be collected from individuals with musculoskeletal problems. Psychometric testing will include test-retest reliability, internal consistency, and construct validity analyses.

The main hypotheses of this study are as follows:

1. The Turkish version of the Generic Functional Index will demonstrate high test-retest reliability when administered to individuals with musculoskeletal disorders.
2. The scores of the Turkish version of the Generic Functional Index will show a significant positive correlation with the scores of the Functional Independence Measure in individuals with musculoskeletal disorders.

DETAILED DESCRIPTION:
Functional assessment is a fundamental component in evaluating the impact of health conditions on individuals' daily lives and in guiding rehabilitation strategies. The Generic Functional Index is a multidimensional instrument developed to assess overall functional status by capturing the effects of a person's problem on their daily activities, mobility, pain, and self-care performance. There is currently no validated Turkish version of the Generic Functional Index available for use in musculoskeletal populations.

This study aims to translate and culturally adapt the Generic Functional Index into Turkish and to investigate its psychometric properties in individuals with musculoskeletal disorders. The adaptation will follow an internationally recognized translation methodology, including forward translation, synthesis, back-translation, expert committee review, and pre-testing. Psychometric evaluation will involve data collection from individuals with musculoskeletal conditions, with analyses focusing on internal consistency, test-retest reliability, and construct validity.

Construct validity will be examined by analyzing the relationship between the Turkish Generic Functional Index and the Functional Independence Measure, which is a widely used tool for assessing independence in daily living activities. A strong correlation between these tools will support the convergent validity of the Turkish Generic Functional Index.

This study is significant because a valid and reliable Turkish version of the Generic Functional Index will provide clinicians and researchers with a standardized tool for evaluating functional limitations in Turkish-speaking populations with musculoskeletal disorders. It will also contribute to the international applicability of the Generic Functional Indexby expanding its use to different cultural and linguistic contexts.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Turkish literacy,
* Cognitive competence,
* Having a musculoskeletal disorder

Exclusion Criteria:

* Those with acute functional impairment
* Those with cognitive impairment, or
* Those with a mental or physical condition that would prevent them from understanding the scale.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with musculoskeletal conditions
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The Turkish Version of Generic Functional Index | T0 and T1 (Baseline and after 1 week after)
  This index is designed for use across a wide range of musculoskeletal and functional conditions and comprises four parts:
  Part 1 - Global Status: Patients rate their overall post-injury status on a 0-10 scale, multiplied by 10 to yield a percentage (range: 0-100).
  Part 2 - Duties and Pain: Assesses functional duties and pain level, each on a 0-10 scale converted to percentages (range: 0-100 each).
  Part 3 - Functional Limitations: A 10-item checklist (mobility, dressing, sleep, etc.), with full or half points; total score (0-10) is multiplied by 10 for a 100-point scale.
  Part 4 - Patient-Specific Index: Patients rate up to 5 activities on a 0-10 scale (0 = worst, 10 = best); total is doubled to yield a percentage (range: 0-100).
  Lower scores indicate greater disability; higher scores reflect better function.
Functional Independence Measure | Baseline
  Functional Independence Measure will be used to examine the construct validity of the Turkish version of the Generic Functional Index. The Functional Independence Measure is a widely accepted and validated tool that assesses functional independence in daily activities through 18 items across motor and cognitive domains, scored on a 7-point scale. Since both instruments aim to evaluate functional status, a significant correlation between Functional Independence Measure and Generic Functional Index scores would support the convergent validity of the Generic Functional Index. Functional Independence Measure's established use in rehabilitation and its robust psychometric properties make it an appropriate reference measure for this validation study. Total Functional Independence Measure scores range from 18 to 126, where lower scores indicate complete dependence and higher scores reflect complete functional independence.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Elcin Dereli, Prof., Study Director — Istanbul Bilgi University; Selina Kara, BSc., Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Beyoglu, Turkey (Türkiye)